CLINICAL TRIAL: NCT02586584
Title: The I-Score Study: The Development and Validation of a Patient-Reported Measure of Antiretroviral Therapy's Interference With Life: A Clinical Patient-management Tool for Healthcare Providers
Brief Title: The I-Score Study: Developing a New Patient-Reported Tool for the Routine HIV Care of Patients on Antiretroviral Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Bertrand Lebouche (Other)
Collaborators: Mitacs (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Bertrand Lebouche, MD, PhD, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: MUHC Study Code 14-229-PSY; Merck-IIS-53538 (Other: Merck Inc); CTN283 (Other: CIHR's Canadian HIV Trials Network)
Record Dates: First submitted 2015-10-20; First posted 2015-10-26 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: HIV/AIDS
Keywords: Patient-Reported Outcome, Antiretroviral Therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this Canada-France study is to develop and validate a multidimensional patient-reported measure of perceived barriers to antiretroviral therapy adherence for HIV-positive patients undergoing treatment that will be theoretically founded, easy to use and helpful to clinicians in their medical decision-making, in a clinical or research setting.

DETAILED DESCRIPTION:
This 24-month study aims to develop and validate a theoretically founded patient-reported outcome measure for use in routine HIV care with patients on antiretroviral therapy (ART). Eight clinical sites will be involved (4 in Canada and 4 in France). The measure will centre on patients' reported barriers to ART adherence and will be adapted for administration via electronic tablet. The study has four main steps. The psychometric validation of the tool and core of the study will be conducted in Step 3. The Observational -Prospective design applies to the field test and retest phase of Step 3. The four steps are nevertheless described below.

Step 1 -Development of the measure's conceptual framework (Start: October 2015)

1. A scoping review of existing HIV-specific patient-reported outcome measures
2. A meta-ethnography of qualitative research on HIV-positive persons' reported barriers to antiretroviral therapy (ART) adherence
3. A content analysis of qualitative interviews with HIV-positive patients on ART about their perceived barriers to adherence (n = 30 patients) The meta-ethnography and content analysis will serve to develop the conceptual framework on which the tool will be based. It will not only define the tool's conceptual domain but outline its relationship to other concepts that will be verified statistically as a part of the tool's validation. Once the framework is completed, the measure will be specified and a bank of items will be generated.

Step 2 -Linguistic validation of the preliminary measure The tool's linguistic validation will involve the professional harmonization of the English and French versions and the creation of a universal French version adapted to all French sites.

Step 3 - Exploration and validation of the measure's psychometric properties

1. During the pilot phase, we will administer our measure and other measures to a small sample size (n = 80) and conduct a number of " cognitive interviews " with participants (n = 8). This will mainly help improve our measure before the field test phase (e.g., by examining missing data, incoherent responses, any problems with question comprehension).
2. The field test (n = 160) will be done with the revised measure of the pilot phase and will include exploratory and confirmatory analyses to examine, among other aspects, the correspondence between the collected data and the conceptual framework developed in Step 1. Here we will also examine the sub-dimensions of our measure and verify the concurrent (e.g., viral load, intention to adhere to ART), convergent (e.g., beliefs about antiretroviral medication) and discriminant (e.g., quality of life) validities of the tool.
3. For the retest phase, the field test participants will be recalled either 1 week or 4 weeks later for another round of data collection to assess the measure's reliability. In this phase an additional measure not included in the previous phase will be included in the questionnaire (adherence to ART). This new measure will be used to verify the predictive validity of the tool.

Step 4 -Pilot the clinical use of the instrument Here, the finalized tool will be applied in a clinical setting with a small sample of HIV-positive patients under ART (n = 24) and their clinicians (n = 8).The aim is to collect data on the tool's perceived utility from the perspective of both populations in order to provide an initial assessment of the feasibility of the tool's wider implementation.

Statistical analyses planned Statistical analyses of the quantitative pilot test phase (n = 80)

* Response coherence
* Analysis of item score distributions
* Analysis of missing data
* Principal components analyses Statistical analyses of the field test phase (n = 160)
* Exploratory analyses
* Confirmatory analyses
* Verification of the measure's convergent, discriminant and concurrent validities Statistical analyses of the retest phase (a random sample of n = 160)
* Principal components analysis and internal consistency through Cronbach's alpha in order to verify whether the factors obtained at the retest phase are the same as those obtained from the field test phase
* Descriptive statistics and multivariate analyses will be carried out in order to compare score means and to verify whether the factors associated with the I-score are the same in phases 2 and 3 Statistical analyses of the Pilot of the instrument's clinical use (n = 24 patients; n = 8 HIV clinicians)
* The statistics produced for this step of the study will be descriptive (e.g., percentages, averages) and comparative. For comparative analyses between patients and their doctors (e.g., on the tool's appreciation), tests will be adapted according to whether the variables used are continuous (e.g., t-tests) or categorical (e.g., chi-square).
* Furthermore, patient and clinician data will be analyzed with a multi-level model to examine, for example, if patient appreciation (or non-appreciation) of the tool is associated or not with differences in the clinicians' perceptions (estimation of individual and structural factors associated with appreciation or non-appreciation).

ELIGIBILITY:
Inclusion Criteria:

* Be a man, woman or transgender person aged 18 years or older
* Be diagnosed HIV-1 positive
* Be treated by a combination of 2 to 3 antiretroviral drugs for at least 3 months
* Ability to speak and understand either French or English

Exclusion Criteria:

* Participation in a clinical trial at the time of enrollment in this study, in some cases (to be discussed on a site-by-site basis by the scientific committee)
* Having a cognitive impairment or medical instability that prevents their use of the electronic tablet, completion of the questionnaire or participation in the interview
* Insufficient mastery of French or English to complete the questionnaires or participate in the interview
* Refusal to use the electronic tablet to fill out the questionnaire material (not relevant for the qualitative and cognitive interviews)
* Co-infection with hepatitis C and currently under treatment for it or having completed hepatitis C treatment 3 months ago or less
* Co-infection with hepatitis B and either not being treated for it or receiving a treatment for it other than one's antiretroviral therapy for HIV
* Participation in the study's Pilot phase (for the field test and retest)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of HIV-positive patients on ART recruited from the caseloads of eight participating clinical sites in France and Canada. The clinical sites were selected on a geographical basis to account for different regional contexts not only in terms of the size of the HIV/AIDS epidemics, but also in terms of the sociodemographic, socioeconomic, and organizational HIV care differences that may exist across regions. The sites are similarly heterogeneous in the representation of risk groups composing the caseloads (e.g., women, injection drug user, men who have sex with men, immigrants).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change in the Interference-Score (I-Score) | During the field test of Step 3 of the study, the I-Score will be administered at week 0 and then at week 4 to evaluate change (reliability)
  The I-Score is the measure to be developed and concerns perceived barriers to antiretroviral therapy adherence

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lebouché, MD PhD, Principal Investigator — McGill University Health Centre, Chronic Viral Illness Service, Royal Victoria Hospital - Glen Site D02.4110 - 1001 boul Décarie, Montreal, QC H4A 3J1
Locations (1):
- Chronic Viral illness Service, Montreal, Quebec, Canada

REFERENCES:
- [Result] Lebouche B, Engler K, Levy JJ, Gilmore N, Spire B, Rozenbaum W, Routy JP. Minimal interference: A basis for selecting ART for prevention with positives. AIDS Care. 2013;25(10):1284-90. doi: 10.1080/09540121.2013.764394. Epub 2013 Feb 11. PMID 23394079
- [Derived] Toupin I, Engler K, Lessard D, Wong L, Lenart A, Spire B, Raffi F, Lebouche B. Developing a patient-reported outcome measure for HIV care on perceived barriers to antiretroviral adherence: assessing the needs of HIV clinicians through qualitative analysis. Qual Life Res. 2018 Feb;27(2):379-388. doi: 10.1007/s11136-017-1711-5. Epub 2017 Oct 13. PMID 29027607